CLINICAL TRIAL: NCT04094753
Title: Think Dry: Optimalisation of Diagnostic Process of Urinary Incontinence in Older People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2013/950
Record Dates: First submitted 2019-08-13; First posted 2019-09-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Incontinence, Urge; Incontinence Stress; Incontinence, Daytime Urinary; Incontinence, Nighttime Urinary
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence, Stress; Diurnal Enuresis; Nocturnal Enuresis | interventions — Blood Specimen Collection; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood Sample — A sober blood sample is taken to observe the following parameters: creatinin, ureum, sodium, potassium, osmolality, HDL cholesterol, LDL cholesterol, triglycerides)
Diagnostic Test: Renal Function Profile — A Renal Function Profile is a 24 hour-urine collection in which urine samples are collected at fixed time points every 3 hours, starting 3 hours after the first morning void. Daytime samples were taken at 10:00-11:30 (U1), 13:00-15:30 (U2), 16:00-17:30 (U3), 19:00-20:30 (U4), and 22:00-23:30 (U5). The nighttime samples were taken at 1:00-2:30 (U6), 4:00-5:30 (U7) and 7:00-8:30 (U8). The volume of each sample, and of each micturition in between, was noted to calculate the 24h, daytime and nighttime urine volume and diuresis rate.
Diagnostic Test: Frequency Volume Chart — Every patient complets a frequency volume chart during 24 of 72 hours
Diagnostic Test: Cystometry — This technique provide the most precise measurement of bladder and urethral sphincter behaviour during bladder filling and during voiding.
Diagnostic Test: Questionaires — Patients have to fulfill the following questionaires
  * ICIQ-Fluts for female participants or ICIQ-Mluts for male participants
  * TILBURG FRAILTY INDICATOR
  * SF-36 Quality of Life score
  * N- QOL
Diagnostic Test: Flow rate measurement + Observation of the post-void residual urine volume — A measurement of the urinary flow rate is observed to collect the maximum Q/s. Afterwards an observation of the PVR is done using ultrasound.
Diagnostic Test: Clinical Examination — Clinical examination of the genital region. For women, coeles are described using the POPQ

SUMMARY:
Urinary incontinence is an increasing medical and socio-economical problem. 44% of the elderly (>65 years) women and 28% of the elderly men suffer from unwilling urine loss. Moreover, this percentages increase with age. Incontinence is a problem with multiple physical, psychological, and financial effects. In addition incontinence has a important impact on the family and healthcare professionals surrounding the elderly.

The problem of urinary incontinence is complex and multifactorial. Moreover, diagnostic guidelines are inconsistent leading to a high amount of technical interventions to diagnose and to specify the type of incontinence.

Aim of this study is to create a short form of necessary technical investigations to diagnose and evaluate urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 years
* Every type of incontinence: stress, urge, mixed.

Exclusion Criteria:

* Patients with an indwelling urinary catheter are doing clean intermittent catheterization are excluded from the study protocol
* Patients with dementia are excluded from the study, based on N-Cog evaluation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older, cognitive intact people (>= 65 years) of both sexes with all types of urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Decreasing the amount of necessary technical investigations to diagnose incontinence | 1 month
  Based on international guidelines different technical investigations are used and approved to observe the type of urinary incontinence individually. Nevertheless, based on expert opinion all technical investigations schould be done together. However this combination of different technical investigations (urodynamics, questionaires, voiding dairy and clinical examination) is not evidence based and time consuming. We want to develop a statistical model to decrease the need of technical investigations to obtain a correct diagnose of stress urinary incontinence, urge urinary incontinence or mixed incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided